CLINICAL TRIAL: NCT04264195
Title: Socially Interactive and Peer Group Regulated Upper Extremity Rehabilitation Following Stroke: Bilateral Activities Compared to Activities With Forced Use of the Paretic Hand (mCIMT) - a Randomized Clinical Trial
Brief Title: Peer Group Regulated mCIMT Program for Adult Stroke Patients: Effects on Functional Activities
Acronym: PEPS-MIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for the Rehabilitation of the Paralysed, Bangladesh (Other)
Collaborators: Jahangirnagar University (Other); Midwestern University (Other); University of Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Fatema Tuj Johra, Principle Investigator,B.Sc. in Occupational Therapy,M.Sc. in Rehabilitation Science, Centre for the Rehabilitation of the Paralysed, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRP.MRS.Iris.2019
Record Dates: First submitted 2020-01-31; First posted 2020-02-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Weakness of Extremities as Sequela of Stroke; Modified Constraint Induced Movement Therapy After Stroke; Upper Extremity Functional Performance After Stroke
Keywords: Stroke; Upper extremity paresis; Recovery of function; Modified CIMT
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: The main element of this model is randomization where participants were randomly assigned into a control group and an experimental group. Both groups got their treatment at the same time for 2 hours for 4 days in a week. The experimental group practiced the tasks with the paretic hand only - the non-paretic hand being constrained by the use of a mitten - where the control group practiced the tasks bimanually.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of Patients: patients are unaware if they are participating in a control or experimental group; groups didn't have contact Masking of investigator: Allocation of patients to treatment group and control group by using sealed envelopes.
  Masking of Assessors: Four assessors (qualified occupational therapists) from both clinical and academic side of CRP were recruited for outcome measurement. Each group had an individual assessor and the same assessor was assigned in pretest, posttest and follow-up assessments. Assessors were not allowed to ask patients for details of the treatment.
  Masking of Therapist: Therapists were randomly allocated into groups before they get (separated) group-specific training in application of the protocol and treatment modality. Therapists have no idea about which is the control group treatment and which is the experimental group treatment. Both groups have got a new, specific way of exercising by a peer regulated group treatment program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-induced movement therapy (Experimental): Constraint-induced movement therapy (PEPS-MIT)
  Interventions: Other: Constraint-induced movement therapy: PEPS-MIT
- Bimanual manipulation (Active Comparator): Bimanual manipulation (PEPS-Bimanual)
  Interventions: Other: Bimanual manipulation exercises (PEPS-Bimanual)

INTERVENTIONS:
Other: Constraint-induced movement therapy: PEPS-MIT — All participants of control and experimental groups received standard stroke rehabilitation. After regular office time, a 2 hours' peer group session was provided, 5 days/week, 4 consecutive weeks, to both groups. One patient 'leads' the group exercises under a therapist's supervision. The therapist is mainly helping and correcting patients during the various exercise tasks.
  • Specific for the experimental group was that patients performed all manipulation tasks with forced use of the paretic hand/arm by wearing a soft-padded mitten at the non-paretic hand, preventing manipulation with that hand. Patients were encouraged to wear the mitten also for 3 hours/day at home, while performing ADL and learned exercises. Behavioural strategies included a treatment contract and daily use of the home activity checklist which was checked by patient's caregiver and signed by both patient and caregiver. Each treatment day the activity checklist was submitted to the therapist who gives feedback.
  Arms: Constraint-induced movement therapy
Other: Bimanual manipulation exercises (PEPS-Bimanual) — All participants of control and experimental groups received standard stroke. After regular office time, a 2 hours' peer group session was provided, 5 days/week, 4 consecutive weeks, to both groups. One patient 'leads' the group exercises under a therapist's supervision. The therapist is mainly helping and correcting patients during the various exercise tasks.
  Specific for the control group was that patients performed all manipulation tasks bimanually, as they used to do in occupational therapy activities. Patients were also asked to document their 'at home' activities in an activity checklist that was regularly checked by the therapists.
  Arms: Bimanual manipulation

SUMMARY:
Each year more than 17 million people in the world are experiencing a stroke. Stroke is a major cause of mortality and one of the prevalent causes of serious disablement.

Stroke sufferers often will have restricted participation in various domains e.g. not being able to fulfill the job requirements. That is why they are losing social contacts and are at risk for social deprivation.

They also show limitations in common daily activities, which implies that they often need help or must use assistive devices because of muscle weakness, spasticity and impaired control over one of the hands, which are very common after stroke. Functional hand recovery will be only minimal at 6 months after stroke in most of the patients. Therefore, patients mainly rely on their unaffected hand to perform daily activities and refrain from using the impaired hand. However, it is known that also after a stroke new connection could be made in the brain when training tasks strenuously. This mechanism is applied in our program by constraint induced movement therapy (CIMT). In CIMT using the unaffected hand is hindered by a mitten, so that patients are forced to perform tasks predominantly with the paretic hand.

The original CIMT protocol includes three main elements:

* Constraining of the non-paretic hand to force the use of paretic hand.
* Repetitive task-oriented training of the paretic hand.
* Adherence-enhancing behavioral methods, to promote the use of this technique in the daily environment.

Although CIMT trials are showing variations in the kind of tasks, the duration of practice per day and the intensity, they all published significant effects of CIMT compared to traditional therapy.

Currently CIMT is worldwide considered the most effective rehabilitation treatment for improving the functioning of the paretic hand in stroke, but this treatment is not applied in Bangladesh. To overcome this,the investigators have made a protocol for CIMT application with the purpose to study the effects in stroke patients in the Bangladesh situation.

Method

Beside the CIMT program the investigators also developed a method for getting maximal social interaction in groups of stroke patients. That may help them to exercise on their own with support of their peers. The investigators call that a 'peer group regulated training' and stroke patients got that training in addition to the usual individually focused rehabilitation. This extra training includes the following elements:

* Stroke patients perform repetitive tasks in a group together (groups 6-8 persons, max 15).
* One of them is assigned as a 'leader', who announces the next task while the therapist is there mainly for helping and correcting patients.
* Tasks are fine-tuned to the Bangladesh' situation regarding gender-specific clothing, manipulation of objects and tasks that needs cognitive solutions.
* Within the training there are socializing tasks like singing, sharing of experiences, complimenting and encouraging each other.
* Patients were asked to perform the tasks by themselves at home as well, and to report about that.

This method was applied in two separate groups. The group that is indicated as the control group mainly performed the exercise tasks bilaterally, as in as usual therapy sessions. The experimental group performed the tasks with forced use of the paretic hand, wearing a mitten at the non-paretic hand.

The investigators will be compared the performances of the two study groups at the start of the group therapy, at the finish one month later, and at 3, 6, 9 and 12 months afterwards.

The hypothesis is that the applied adherence-enhancing behavioral method will have dominant effects, and that the methods: 'bilaterally' versus 'forced use of paretic arm/hand' (CIMT) will show equal improvements in the short and longer term.

DETAILED DESCRIPTION:
Research Question. To compare the performances of the experimental and control groups at the start of the PEPS program, at the finish 1 month later and at 3, 6, 9 and 12 months follow up.

Hypothesis. Null Hypothesis H0: µ1- µ2 = 0 or μ1=μ2; where μ1= mean of experimental group and μ2= mean of control group.

PEPS-MIT is not more effective than PEPS-bimanual training in Restoration of upper limb functioning following stroke.

Alternative Hypothesis Ha: µ1- µ2> 0 or µ1> µ2 PEPS-MIT is more effective than PEPS-bimanual training in Restoration of upper limb functioning following stroke.

Ethical Considerations. The Bangladesh Health Professions Institute Institutional Review Board (IRB) judged the ethical issues and they gave the permission for data collection. All data and assessment files were stored in security and files were maintained with patient data held anonymously.

All patients were given information about the trial and they were secured that withdrawing from the trial didn't give any consequences for their normal treatment. All eligible patients wish to participate and they all signed informed consent forms.

Study design. The study is a double blind randomized clinical trial with baseline assessment, post-treatment assessment and three-month, 6 months, 9 months and 12 months follow-up, two group comparison design.

Sample Size. The study sample was all the CRP rehabilitation center patients who meet the inclusion criteria within the study time frame (10.08.18 to 25.12.18). Total 140 patients meet the criteria, and all are allocated to the study. Through simple random techniques patients were allocated into control group and experimental group according to a 1:1 ratio. Thus, after randomization 70 patient were allocated into control group and 70 were allocated into experimental group. Sealed envelope was used for randomization that was carried out by the director of the Spinal Cord Injury Rehabilitation unit of Occupational Therapy Department. Patients are blinded for the therapy group.

Interventions. The fundamental PEPS-method (Please see PEPS training programme full description, URL link- https://www.crp-bangladesh.org/standard-treatment-program) was applied in both the control and experimental group.

The control group mainly performed the exercise tasks bimanually, as in as usual' therapy sessions (PEPS-bimanual), whereas the experimental group performed the exercise tasks with forced use of the most affected hand (wearing a specially designed mitten at the non-paretic hand; PEPS-MIT).

Treatment sessions. Two hours in 5 days per week; Total 4 weeks. Assessments. Trained assessors who were blinded for the intervention had assessed the functioning of the upper limb before the start of the treatment, at the end and at follow-up after 3, 6, 9 and 12 months.

Therapists. Therapists were only facilitator of the peer lead training sessions. Six qualified therapists were randomly (through sealed envelope) allocated to either the experimental or the control group. Therapists of both groups have got a 7 days training in the core PEPS program. Both groups of therapists were forbidden to share their training knowledge with each other as part of study protocol. Therapists are unaware which group is the control and which is the experimental group: they were blinded for the intervention.

Quality assurance. Pilot trial: Investigators conducted a pilot trial (20 days with 4 patients) before conducting the study for checking feasibility of the program and outcome measures.

Each session therapist asked the patients for experiencing adverse events, and registered these.

Monitoring the process of training and data registration regarding the home-exercising was done during three days each week by the first and third author.

The statistics department of Jahangirnagor University (JU) and MRS program, BHPI, CRP helps in site monitoring and auditing, and in controlling the accuracy and completeness of the data, in data validation and registry procedure. All data were checked by Statistics department of JU and rechecked by MRS program, BHPI, CRP.

Investigators have made a log-book with descriptions of each variable and the normal range of scores per test, and the codes to indicate the individual patients to keep the patient data anonymously.

All data were put into SPSS files and checked. Missing data. There are no missing data in initial assessments.For missing data in follow-up assessments (no show of patients, or because of passing away of patients) will be used the 'intention-to-treat' analysis.

Statistical analysis: 1. Independent t tests and Chi- Square (χ2) tests will be used to compare the control and experimental group on sociodemographic and disease variables. Changes in test scores within each group were evaluated with paired t tests, and between groups with independent t-test. Repeated measure ANOVA (factorial ANOVA) model will be used to see whether group differences existed or not and how group scores changes over time and interaction between Group*Time.

ELIGIBILITY:
Inclusion Criteria:

* Acute (four weeks- three months) to chronic (above three months to one year) stage post stroke patients.
* Diagnosis of a first stroke.
* Unilateral hand impairment.
* Must have more than 10 to 20 degrees active wrist extension and 10 degrees active finger extension.
* Having 20 points or more on the Mini-Mental State Examination scale.
* Age range 18-75 years and first stroke.
* Willing to participate in the study and signed the informed consent form.

Exclusion Criteria:

* Persons with other neurological disorders.
* Bilateral stroke.
* Recurrent stroke history.
* Unstable cardiovascular diseases is excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test - Functional Ability (WMFT-FA) | Changes between score from pre-treatment, immediately post-treatment and at 3, 6, 9 and 12 months follow-up.
  The WMFT-FA consists of 15 timed arm movement tasks (outcomes in seconds; maximum time to complete a task:120 sec.) plus 2 strength tasks (outcomes in lbs and kg(s) lifted). All items are scored on a six point functional ability scale (minimum score is 0 and maximum score is 5 ).

SECONDARY OUTCOMES:
Nine Holes Peg Test (NHPT) | Changes between score from pre-treatment, immediately post-treatment and at 3, 6, 9 and 12 months follow-up.
  The Nine Holes Peg Test (NHPT) is a dexterity measure for the upper extremities. A stopwatch was used to measure the time taken to place the 9 pegs in wooden hole pegboard.
Action Research Arm Test (ARAT) | Changes between score from pre-treatment, immediately post-treatment and at 3, 6, 9 and 12 months follow-up.
  Action Research Arm Test (ARAT) is a quantitative test for upper extremity Function. There are four subsets: Grasp, GRIP, Pinch and Gross arm movement with each item graded on a 4-point ordinal scale for a total possible score of 57.
Motor activity Log scale (MAL) | Changes between score from post-treatment and at 3, 6, 9 and 12 months follow-up.
  The Motor Activity Log Scale (MAL) is a structured interview comprising 30 standardized questions encompassing various ADL tasks, which was used to assess the subjects' subjective report of 30 common daily tasks. It included two assessment subscales that rate the more affected upper extremity regarding the amount of use (AOU) and the quality of movement (QOM) .
Fugl -Meyer assessment (FMA-Upper Extremity Motor Section) | Changes between score from pre-treatment, immediately post-treatment and at 3, 6, 9 and 12 months follow-up.
  The FMA is used to measure motor impairment. The upper-extremity motor part includes 33 items scored on a 3-point ordinal scale for a possible minimum score is 0 and maximum is 66.
Functional Independence measure (FIM: Self-care Section) | Changes between score from pre-treatment, immediately post-treatment and at 3, 6, 9 and 12 months follow-up.
  The Functional Independence FIM-Self care section has 7 items that objectively measures changes in basic ADL function ( minimum score is 1 and maximum is 59).

CONTACTS AND LOCATIONS:
Overall Officials: Fatema Tuj Johra, M.Sc., Principal Investigator — Centre for the Rehabilitation of the Paralysed; Clara Dorothea (Dorine) Van Ravensberg, PhD, Study Chair — Centre for the Rehabilitation of the Paralysed; Md. Forhad Hossain, PhD, Study Chair — Department of Statistics, Jahangirnagar University, Bangladesh; Mark Kovic, PhD, Study Chair — Associate Program Director,Occupational Therapy Department,Midwestern University ,USA
Locations (1):
- Centre for the Rehabilitation of the Paralysed, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Study protocol,Statistical Analysis Plan,Clinical Study Report will be share after trial result publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 10 months after trial result publication till 1 year later.
Access Criteria: Researchers having already published studies in stroke and CIMT trials. For secondary analyses of data,preferably for eligibility and predictive outcome model for the peer regulated group exercise program (PEPS) and the PEPS-MIT intervention.
  Requests will be reviewed by the principle investigator and facility contact person.

REFERENCES:
- See also: PEPS training programme full description — https://www.crp-bangladesh.org/standard-treatment-program
- See also: PEPS training programme full description — http://www.bhpi.edu.bd/standard-treatment-program/